CLINICAL TRIAL: NCT04082208
Title: Use of High Flow Nasal Cannula in Patients Undergoing Endoscopic Retrograde Cholangiopancreatography (ERCP) Under Sedation. Comparative, Randomized Study of Two Health Products Approved by the Community
Brief Title: High Flow Nasal Cannula in Patients Undergoing Endoscopic Retrograde Cholangiopancreatography (ERCP) HF-study
Acronym: HFS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, JULIA MARTÍNEZ OCÓN, Anesthesiologist, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: High-Flow study-172
Record Dates: First submitted 2019-09-04; First posted 2019-09-09 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Patient Population Submitted to ERCP
Keywords: ERCP; High Flow nasal cannula; deep sedation

STUDY DESIGN:
Intervention Model Description: Unicentre controlled clinical trial, unmasked, performed in the Digestive Endoscopy Unit of the Hospital Clínic. 172 patients submitted to Endoscopic Retrograde Cholangiography who agree to participate in the study will be included consecutively and randomly.
  Patients will be randomized into two groups: Control group: low flow device (nasal glasses) and High Flow device group (LAF).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): High Flow nasal cannula (HF)
  Interventions: Device: High Flow nasal cannula
- Standar Care Group (Active Comparator): Standar Care: low flow device (LF)
  Interventions: Device: Low Flow nasal cannula

INTERVENTIONS:
Device: High Flow nasal cannula — Administration of high flow nasal cannula during ERCP procedure
  Arms: Intervention Group
Device: Low Flow nasal cannula — Administration of low flow nasal cannula during ERCP procedure: standard care
  Arms: Standar Care Group

SUMMARY:
The expected results with this study are that high flow devices (LAF) provide adequate respiratory support during the performance of ERCP under deep sedation, reducing episodes of desaturation, hypoventilation and airway obstruction compared to low flow devices ( nasal glasses).

DETAILED DESCRIPTION:
Deep sedation performed during the ERCP technique associates an increased risk of decrease in Sat02%, hypercapnia and airway obstruction with consequences ranging from interruption or suspension of the technique to complications that may put the patient's life at risk .

High flow devices (HF) due to the pressurization capacity of the airway and the reduction of anatomical dead space will favor a better gas exchange compared to low flow devices (LF), which will manifest clinically with a reduction in episodes of decrease of Sat02% and a decrease in carbon dioxide levels.

The main objective of the study is to demonstrate that the use of high flow devices (HF) decreases the episodes of desaturation (defined as Sat02 ≤ 90% measured through pulse oximetry) that occur during the performance of ERCP under deep sedation compared to Low flow devices (LF) with equal Inspiratory oxygen fraction (Fi02) in both cases.

The expected results with this study are that high flow devices (LAF) provide adequate respiratory support during the performance of ERCP under deep sedation, reducing episodes of desaturation, hypoventilation and airway obstruction compared to low flow devices ( nasal glasses).

ELIGIBILITY:
Inclusion Criteria:

* Patients Age over ≥18 years. Willing to participate

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Desaturation during ERCP | 2 years
  Demonstrate that the use of high flow devices (HF) decreases episodes of desaturation (defined as Sat02 ≤ 90% measured by pulse oximetry) that occur during the performance of ERCP under deep sedation compared to low flow devices ( LF).

SECONDARY OUTCOMES:
CO2 during ERCP | 2 years
  The use of HF decreases the CO2 levels measured through transcutaneous CO2 (PtcCO2) compared to conventional oxygen therapy (LF)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Martinez Ocon, Dr, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Clinic Hospital (Endoscopy Unit), Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No